CLINICAL TRIAL: NCT02860325
Title: Non-invasive Neurally Adjusted Ventilatory Assist Versus nCPAP or Non Synchronized NIPPV in Preterm Infants Under 32 Weeks Gestational Age: A Randomized Clinical Trial
Brief Title: NIV-NAVA Versus Nasal Continuous Positive Airway Pressure (nCPAP) or Non Synchronized NIPPV
Acronym: Bio-NAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario Universitario Insular Materno Infantil (Other)
Responsible Party: Principal Investigator, Fermín García-Muñoz Rodrigo, Head of Neonatal Unit, Complejo Hospitalario Universitario Insular Materno Infantil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC-CHUIMI-2014/761
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Respiratory Distress Syndrome, Newborn; Apnea of Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIV-NAVA (Experimental): Patients allocated to non-invasive NAVA
  Interventions: Device: NIV-NAVA
- Conventional (Active Comparator): Patients allocated to nasal CPAP or non-synchronized nasal IPPV
  Interventions: Device: Conventional

INTERVENTIONS:
Device: NIV-NAVA — Non-invasive ventilatory support by means of neurally adjusted ventilatory assist (SERVO-n, Maquet, Solna, Sweden)
  Arms: NIV-NAVA
Device: Conventional — Non-invasive ventilatory support by means of nCPAP or non-synchronized nIPPV (Infant Flow, CareFusion)
  Arms: Conventional

SUMMARY:
Mechanical respiratory support of preterm neonates with respiratory distress syndrome (RDS) and/or apnoea of prematurity (AOP) might be associated with adverse effects due to positive pressure (barotrauma), excessive gas delivery (volutrauma) or inadequate volume (atelectrauma). Asynchrony between patient efforts and ventilator support increases patient discomfort, favouring "fighting" the machine, and increases the risk of air trapping and lung overdistension even in patients with non-invasive ventilation (NIV).

Recently, a new modality of synchronization has been available for pediatric and neonatal use: the neurally adjusted ventilatory assist (NAVA), which uses the diaphragmatic electrical activity (Edi) as a signal to start the rise in pressure of the ventilator, and to adjust the tidal volume and the inspiratory time (cycling off) to the patient needs, breath by breath.

The aims of this study are to know whether NIV-NAVA compared to unsynchronized modalities (nCPAP/nIPPV), in infants born < 32 weeks GA with respiratory distress syndrome or requiring prophylactic NIV (immaturity, apnoea) reduces systemic inflammation, measured by serum cytokines concentration, reduces the need for oxygen and respiratory support, and if it increases the probabilities of survival without bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
Introduction. Mechanical respiratory support of preterm neonates with respiratory distress syndrome (RDS) and/or apnoea of prematurity (AOP) might be associated with adverse effects as a consequence of positive pressure use (barotrauma), excessive gas delivery (volutrauma) or inadequate volume (atelectrauma). All these factors could give rise to an increase in the alveolo-capillary membrane permeability, alveoli oedema, hyaline membrane formation and epithelial cells desquamation. These phenomena eventually could lead to activation of inflammatory mediators (biotrauma) with local and systemic noxious effects.

During assisted ventilation, the lack of synchrony between patient efforts and ventilator support increases patient discomfort, favouring "fighting" the machine, and increases the risk of air trapping and lung overdistension. Even in patients with non-invasive ventilation (NIV), uneasiness and respiratory distress would cause air hunger, developing intrapleural negative pressure with risk of lung overinflation despite using low airway positive pressures. The use of neuromuscular blockade in adults with acute respiratory distress syndrome (ARDS) has been associated with a decrease in serum cytokine levels and 90 days adjusted mortality.

NAVA uses the diaphragmatic electrical activity (Edi) as a signal to start the rise in pressure of the ventilator. Likewise, it allows automatic adjustment of peak inspiratory pressure (PIP) to the patient's effort, providing variable tidal volume according to his/her needs. Finally, the system allows the inspiratory cycling off with Edi decline (normally set at 70% of Edi Peak), that is, with diaphragmatic relaxation. NAVA has shown a faster response time and a better level of synchronization than traditional flow or pressure systems, achieving greater comfort levels in adults and paediatric patients. Some paediatric and neonatal studies have shown a reduction in PIP, without changes in mean airway pressure (MAP), and a reduction in oxygen requirement (FiO2). These changes were not associated with major complications (intraventricular haemorrhage, pneumothorax, or necrotizing enterocolitis).

A relevant target in neonatal ventilatory support is to minimize the aggression to the lungs and respiratory system using NIV whenever possible, and/or extubating patients as soon as possible. For this reason, profound sedation, analgesia, or neuromuscular blockade are rarely indicated in the newborn period. NAVA synchronization might improve patient comfort, preventing patient-ventilator fighting, and lung overinflation episodes (volutrauma), ultimately reducing biotrauma. To the knowledge of the investigators, studies evaluating this new ventilatory modality (NAVA) in the newborn period are still scarce, and its potential to reduce inflammation has not been tested.

Objectives.

To determine if NIV-NAVA compared to unsynchronized modalities (nCPAP/nIPPV), in infants born < 32 weeks GA with respiratory distress syndrome or requiring prophylactic NIV (immaturity, apnoea):

1. Reduces systemic inflammation, measured by serum cytokines concentration.
2. Reduces the need for oxygen and respiratory support.
3. Increases the probabilities of survival without bronchopulmonary dysplasia (BPD).

Design. Single centre, prospective and controlled randomized clinical trial.

Setting. Tertiary Hospital with near 6000 births per year and a Neonatal Intensive Care Unit (NICU) with 15 beds and approximately 250 admissions per year.

Methods. Informed consent (IC) will be obtained before birth, during mothers' admission with threatened preterm labour. Once the IC is obtained and after the infant's birth, patients will be randomized by a random numbers table, kept in sealed envelops, to "Group A" (NAVA) or "Group B" (conventional strategies).

In all cases meeting inclusion criteria, a cord blood sample will be collected to determine the level of cytokines: Tumour necrosis factor alpha (TNF - α), interleukin (IL) 1 beta (IL-1ß), IL-6, and IL-8.

The decision to intubate in delivery room or to provide NIV will be carried out by the attending neonatologist at time of birth based on clinical criteria. In our unit, standard care is intubation and prophylactic surfactant administration in delivery room in neonates < 25 weeks GA, or older babies that did not received antenatal steroid and need intubation during resuscitation. Neonates 26 - 29 weeks GA with adequate respiratory effort are resuscitated and transferred to NICU with NIV (Neo-puff ®). Preterm babies > 29 weeks GA receive respiratory support (invasive or NIV) only when clinically indicated.

After admission to NICU, patients requiring invasive mechanical ventilation will be supported according to theirs needs and the criteria of the attending neonatologist. In our unit, modes with volume guarantee (VG) or volume control are currently used: Assist/Control+VG, Synchronized - Intermittent Mandatory Ventilation (S-IMV)+VG, and Pressure Regulated Volume Control (PRVC). After extubation and in patients supported non-invasively since the beginning, NIV will be provided according to randomization group:

Group A: With the ventilator SERVO-n (Maquet, Solna, Sweden), in NIV-NAVA mode. The ventilation parameters (PEEP, FiO2, NAVA level, etc.) will be established and adjusted by the attending clinician according to the patient's needs.

Group B: With the Infant Flow device (CareFusion) in nCPAP or non-synchronised Biphasic mode. The ventilation parameters (Flow, PEEP, FiO2, PIP level, etc.) will be established and adjusted by the attending clinician according to the patient's needs.

Surfactant (Curosurf ®, 100 mg/kg) will be administered according to clinical indications following the Unit's protocol. In general, if the patient did not receive it in delivery room, it is administered as soon as possible in the NICU when the patient needs FiO2 >0.3. Intubated patients will receive surfactant through a double lumen tube, and those with NIV by a minimally invasive method, or by the Insure (intubate, surfactant, and extubated) method.

Quantitative cytokine determination will be carried out simultaneously in all samples by X-MAP technology using the Bioplex cytometer (Biorad) which allows the simultaneous measure of multiple analytes.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns < 32 weeks GA with neonatal respiratory distress syndrome, diagnosed by clinical and radiological findings who need invasive or non-invasive mechanical ventilation.
2. Newborns < 29 weeks of gestation (GA) with non-invasive mechanical ventilation at admission indicated as per protocol.
3. Previous parent or legal guardian authorization (informed consent).

Exclusion Criteria:

1. Major congenital malformation or chromosomal abnormality.
2. Absence of informed consent.
3. Outborn patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Survival without moderate or severe bronchopulmonary dysplasia (BPD) | From admission to first discharge from hospital, assessed up to 1 year
  Moderate or severe BPD: dependency on supplemental oxygen and/or ventilatory support at 36 weeks postmenstrual age (PMA) or at hospital discharge (what happens first).

SECONDARY OUTCOMES:
Blood level of cytokines: Tumor necrosis factor alpha (TNF-α), interleukin (IL) 1 beta (IL-1ß), IL-6, and IL-8. | T-0: cord blood or immediately after admission; T-1: 48 to 72 h.; T-2: 5th to 7th day of life; and T-3: 28th day of life.
  Level of the different cytokines in blood
Total time of ventilatory support (in days) | From admission to first discharge from hospital, assessed up to 1 year
  Number of days with invasive and/or non-invasive ventilatory support
Intervention failure | From admission to first discharge from hospital, assessed up to 1 year
  Need for intubation
Total time of oxygen therapy (in days) | From admission to first discharge from hospital, assessed up to 1 year
  Numer of days with supplementary oxygen
Length of stay (in days) | From admission to first discharge from hospital, assessed up to 1 year
  Number of days in hospital until first discharge

OTHER OUTCOMES:
Intraventricular haemorrhage (IVH) and grade | From admission to first discharge from hospital, assessed up to 1 year
  According to Papile's classification
Periventricular leukomalacia (PVL) | From admission to first discharge from hospital, assessed up to 1 year
  Cysts or hyperecogenicities for more tan 14 days
Retinopathy of Prematurity (ROP) stage and need for laser therapy | From admission to first discharge from hospital, assessed up to 1 year
  Grade 3 or higher (International classification).
Necrotizing Enterocolitis (NEC) and stage | From admission to first discharge from hospital, assessed up to 1 year
  Grade 2 or greater of Bell's classification

CONTACTS AND LOCATIONS:
Overall Officials: Fermín García-Muñoz Rodrigo, Ph.D, Principal Investigator — Head of Neonatal Unit
Locations (1):
- Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tremblay LN, Slutsky AS. Ventilator-induced injury: from barotrauma to biotrauma. Proc Assoc Am Physicians. 1998 Nov-Dec;110(6):482-8. PMID 9824530
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Stein H, Firestone K, Rimensberger PC. Synchronized mechanical ventilation using electrical activity of the diaphragm in neonates. Clin Perinatol. 2012 Sep;39(3):525-42. doi: 10.1016/j.clp.2012.06.004. PMID 22954267
- [Result] Forel JM, Roch A, Marin V, Michelet P, Demory D, Blache JL, Perrin G, Gainnier M, Bongrand P, Papazian L. Neuromuscular blocking agents decrease inflammatory response in patients presenting with acute respiratory distress syndrome. Crit Care Med. 2006 Nov;34(11):2749-57. doi: 10.1097/01.CCM.0000239435.87433.0D. PMID 16932229
- [Result] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Result] de la Oliva P, Schuffelmann C, Gomez-Zamora A, Villar J, Kacmarek RM. Asynchrony, neural drive, ventilatory variability and COMFORT: NAVA versus pressure support in pediatric patients. A non-randomized cross-over trial. Intensive Care Med. 2012 May;38(5):838-46. doi: 10.1007/s00134-012-2535-y. Epub 2012 Apr 6. PMID 22481227
- [Result] Breatnach C, Conlon NP, Stack M, Healy M, O'Hare BP. A prospective crossover comparison of neurally adjusted ventilatory assist and pressure-support ventilation in a pediatric and neonatal intensive care unit population. Pediatr Crit Care Med. 2010 Jan;11(1):7-11. doi: 10.1097/PCC.0b013e3181b0630f. PMID 19593246
- [Result] Stein H, Howard D. Neurally adjusted ventilatory assist in neonates weighing <1500 grams: a retrospective analysis. J Pediatr. 2012 May;160(5):786-9.e1. doi: 10.1016/j.jpeds.2011.10.014. Epub 2011 Dec 3. PMID 22137670